CLINICAL TRIAL: NCT03166605
Title: Ingestion of Simethicone After Capsule Ingestion and Its Impact on Quality of Video Capsule Endoscopy- a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Gurjiwan Virk, MD, Resident Physician, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4849
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Video Capsule Endoscopy
MeSH Terms: interventions — Simethicone

STUDY DESIGN:
Intervention Model Description: Control, Sham , Experimental
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): First group: Control
  Follow the current standard protocol used at Albany Medical Center that includes:
  * Do not drink anything for an additional 2 hours after swallowing pill cam. After which patient may drink clear liquids
  * Do not eat solid food until 4 hours after swallowing. After which patient may eat light that includes soup, toast.
  * Return to clinic (RTC) 8 hours after to remove equipment
  * Avoid carbonated beverages and gas forming foods for the completion of the 8-hours study period
- Sham (Sham Comparator): * Receive 3 ml simethicone 20 minutes prior to capsule swallowing
  * Do not drink anything for an additional 2 hours after swallowing pill cam. After which patient may drink clear liquids
  * Do not eat solid food until 4 hours after swallowing. After which patient may eat light that includes soup, toast.
  * Return to clinic (RTC) 8 hours after to remove equipment
  * Avoid carbonated beverages and gas forming foods for the completion of the 8-hours study period.
  Interventions: Drug: Simethicone
- Experiment (Experimental): * Receive 3 ml simethicone 20 minutes prior to capsule swallowing.
  * Receive 3 ml simethicone 1 hours after capsule swallowing
  * Receive 1.5 ml simethicone 2 hours after capsule swallowing
  * Do not drink anything for an additional 1 hour after taking last simethicone dose. After which patient may drink clear liquids
  * Do not eat solid food until 4 hours after swallowing. After which patient may eat light that includes soup, toast.
  * Return to clinic (RTC) 8 hours after to remove equipment
  * Avoid carbonated beverages and gas forming foods for the completion of the 8-hours study period.
  Interventions: Drug: Simethicone

INTERVENTIONS:
Drug: Simethicone — Giving simethicone before and after capsule ingestion.
  Arms: Experiment; Sham

SUMMARY:
Wireless video capsule endoscopy (VCE) is a non-invasive technology that looks into small intestine and gives images of its lumen as the wireless capsule passes through it. It is used widely to access this anatomically difficult part of the body that cannot be seen via either colonoscopy or endoscopy. Currently various studies have been done that give multiple comparisons between various bowel preparation in terms of quality of the small bowel visualization. No studies have been done where simethicone (Gas-X) is ingested after capsule swallowing. We intend to give patients simethicone 1 hour after capsule ingestion for two consecutive hours and compare results of capsule endoscopy outcomes like small bowel transit time (SBTT), diagnostic yield (DY), small bowel visualization quality (SBVQ) and completion rate (CR).

DETAILED DESCRIPTION:
Currently various studies have been done that give multiple comparisons between various bowel preparation in terms of small bowel transit time (SBTT), diagnostic yield (DY), small bowel visualization quality (SBVQ), completion rate (CR). Studies suggest that using Polyethylene glycol (PEG) prep is significantly better compared to clear liquid and overnight fast in terms if SBVQ and DY (Rokkas et al 2009). Other studies have shown using simethicone 30 minutes before capsule ingestion increases visibility compared to clear liquid and PEG preparation but no significant difference in gastrointestinal transit time or examination completion rate (Wei et al 2008). No studies have been done where simethicone is ingested after capsule swallowing.

Simethicone helps absorb the air bubble in the lumen which can improve the image quality. It decreases the surface tension of gas bubbles thereby dissolving them and preventing gas pockets from forming in GI system. It's often used over the counter for gas relief. Gastric emptying time is usually less than 5 hours, small bowel transit time is usually less than 6 hours, and colonic transit time is usually less than 59 hours (Rao et al 2009). Giving simethicone till 2 hours after swallowing capsule can help clear gas bubble before the capsule migrates into the small bowel.

Albert et al 2004 gave patients 80mg simethicone before swallowing the wireless capsule for their study. Wei et al 2008 gave 300mg of simethicone 20 minutes before swallowing the capsule. Chen et al 2011 gave 20ml (40mg/ml) simethicone 30 minutes before capsule ingestion which amounts to 800 mg total. Current FDA recommendation for adults is 500mg maximum daily dose. The liquid form comes in concentration of 20mg/0.3ml which constitutes to 7.5 ml for 500mg dose.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 and older
* patients undergoing capsule endoscopy for standard of care
* patients able to give consent for themselves

Exclusion Criteria:

• prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Small bowel visualization quality (SBVQ) | 8 hours

SECONDARY OUTCOMES:
Small bowel transit time (SBTT), | 8 hours
Diagnostic yield (DY) | 8 hours
completion rate (CR) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Asra Batool, MD, Principal Investigator — Albany Medical College; Gurjiwan s Virk, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany medical center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Does purgative preparation influence the diagnostic yield of small bowel video capsule endoscopy?: A meta-analysis. Rokkas T, Papaxoinis K, Triantafyllou K, Pistiolas D, Ladas SD Am J Gastroenterol. 2009;104(1):219. Purgative bowel cleansing combined with simethicone improves capsule endoscopy imaging. Wei W, Ge ZZ, Lu H, Gao YJ, Hu YB, Xiao SD Am J Gastroenterol. 2008;103(1):77. Investigation of colonic and whole-gut transit with wireless motility capsule and radiopaque markers in constipation.Rao SS, Kuo B, McCallum RW, Chey WD, DiBaise JK, Hasler WL, Koch KL, Lackner JM, Miller C, Saad R, Semler JR, Sitrin MD, Wilding GE, Parkman HP Clin Gastroenterol Hepatol. 2009;7(5):537. Optimal Bowel Preparation for Video Capsule Endoscopy. Hyun Joo Song, Jeong Seop Moon, and Ki-Nam Shim. Gastroenterology Research and Practice, vol. 2016, Article ID 6802810, 7 pages, 2016. doi:10.1155/2016/6802810 Simethicone for small bowel preparation for capsule endoscopy: a systematic, single-blinded, controlled study. Albert J, Göbel CM, Lesske J, Lotterer E, Nietsch H, Fleig WE Gastrointest Endosc. 2004;59(4):487 Small bowel preparations for capsule endoscopy with mannitol and simethicone: a prospective, randomized, clinical trial. Chen HB, Huang Y, Chen SY, Song HW, Li XL, Dai DL, Xie JT, He S, Zhao YY, Huang C, Zhang SJ, Yang LN J Clin Gastroenterol. 2011;45(4):337.
- [Result] Wei W, Ge ZZ, Lu H, Gao YJ, Hu YB, Xiao SD. Purgative bowel cleansing combined with simethicone improves capsule endoscopy imaging. Am J Gastroenterol. 2008 Jan;103(1):77-82. doi: 10.1111/j.1572-0241.2007.01633.x. Epub 2007 Nov 15. PMID 18005366
- [Result] Rao SS, Kuo B, McCallum RW, Chey WD, DiBaise JK, Hasler WL, Koch KL, Lackner JM, Miller C, Saad R, Semler JR, Sitrin MD, Wilding GE, Parkman HP. Investigation of colonic and whole-gut transit with wireless motility capsule and radiopaque markers in constipation. Clin Gastroenterol Hepatol. 2009 May;7(5):537-44. doi: 10.1016/j.cgh.2009.01.017. PMID 19418602
- [Result] Song HJ, Moon JS, Shim KN. Optimal Bowel Preparation for Video Capsule Endoscopy. Gastroenterol Res Pract. 2016;2016:6802810. doi: 10.1155/2016/6802810. Epub 2015 Dec 31. PMID 26880894
- [Result] Albert J, Gobel CM, Lesske J, Lotterer E, Nietsch H, Fleig WE. Simethicone for small bowel preparation for capsule endoscopy: a systematic, single-blinded, controlled study. Gastrointest Endosc. 2004 Apr;59(4):487-91. doi: 10.1016/s0016-5107(04)00003-3. PMID 15044883
- [Result] Chen HB, Huang Y, Chen SY, Song HW, Li XL, Dai DL, Xie JT, He S, Zhao YY, Huang C, Zhang SJ, Yang LN. Small bowel preparations for capsule endoscopy with mannitol and simethicone: a prospective, randomized, clinical trial. J Clin Gastroenterol. 2011 Apr;45(4):337-41. doi: 10.1097/MCG.0b013e3181f0f3a3. PMID 20871410